CLINICAL TRIAL: NCT05179954
Title: Apolipoprotein C3-loading of Apolipoprotein B100 Lipoproteins and Cardiovascular Disease in Patients With Type 1 Diabetes
Brief Title: Lipoprotein Kinetics in T1D
Acronym: LTD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Bettina Mittendorfer, Senior Associate Dean for Research, University of Missouri-Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2097324
Record Dates: First submitted 2021-11-22; First posted 2022-01-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Comprehensive Metabolic Panel

STUDY DESIGN:
Intervention Model Description: Cross-sectional comparison (T1D vs healthy control)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Healthy control group
  Interventions: Other: Metabolic testing
- T1D group (Active Comparator): T1D group
  Interventions: Other: Metabolic testing

INTERVENTIONS:
Other: Metabolic testing — Participants will complete a metabolic testing protocol that includes intravenous infusion of stable isotope labeled tracers and blood sampling to determine lipoprotein kinetics

SUMMARY:
The purpose of this research study is to understand how type 1 diabetes (T1D) increases the risk for cardiovascular diseases (heart attack and stroke). To this end, the investigators will compare apolipoprotein and triglyceride kinetics in people wtih T1D and healthy control participants.

DETAILED DESCRIPTION:
Not required

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 but ≤45 years
* premenopausal/eumenorrheic and not pregnant or breastfeeding
* non-obese (body mass index ≥18.5<30.0 kg/m2)
* Fasting plasma triglyceride <150 mg/dL

Additional inclusion criteria for control subjects:

* Fasting plasma glucose <100 mg/dL
* Plasma glucose 2 h after a 75 g oral glucose challenge <140 mg/dL
* HbA1c <5.6%.

Additional inclusion criteria for subjects with T1DM:

* stable insulin regimen (multiple daily insulin injections or continuous subcutaneous insulin) for at least 8 weeks before screening
* no use of diabetes medications other than insulin
* HbA1c <8.0%, basal (overnight fasted)
* no severe symptomatic hypoglycemic event associated with a seizure or requiring help from other people or a medical facility in the 6 months prior to screening or metabolic testing

Exclusion Criteria:

* more than 1.5 h of structured exercise/week
* use of tobacco products, excessive amounts of alcohol, or dietary supplements and/or medications known to affect lipid metabolism
* hypothyroidism or other disorders known to affect lipid metabolism
* conditions that would make it impossible to complete the study protocol

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Apolipoprotein C turnover rate | one time, at baseline (this is a cross-sectional, observational study, no intervention)
  Apolipoprotein C turnover rate will be assessed by using an intravenous stable isotope labeled amino acid infusion

SECONDARY OUTCOMES:
Triglyceride turnover rate | one time, at baseline (this is a cross-sectional, observational study, no intervention)
  Triglyceride turnover rate will be assessed by using an intravenous stable isotope labeled glycerol infusion
Apolipoprotein B-100 turnover rate | one time, at baseline (this is a cross-sectional, observational study, no intervention)
  Apolipoprotein B-100 turnover rate will be assessed by using an intravenous stable isotope labeled amino acid infusion
Apolipoprotein C concentration | one time, at baseline (this is a cross-sectional, observational study, no intervention)
  Apolipoprotein C concentration
Triglyceride concentration | one time, at baseline (this is a cross-sectional, observational study, no intervention)
  Triglyceride concentration
Apolipoprotein B-100 concentration | one time, at baseline (this is a cross-sectional, observational study, no intervention)
  Apolipoprotein B-100 concentration

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Mittendorfer, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri School of Medicine, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be available upon reasonable request
Time Frame: 5 years after completion of the study